CLINICAL TRIAL: NCT05216393
Title: RecTech Match Feasibility Testing (RERC on Exercise and Recreational Technologies for People With Disabilities- RECTECH IV)
Brief Title: A Person-Centered Geotagged Social Networking System to Promote Physical Activity in the Community
Acronym: RECTECHIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mohanraj Thirumalai, assistant professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 300007761
Record Dates: First submitted 2021-12-16; First posted 2022-01-31 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Physical Inactivity; Disability Physical
Keywords: physical activity; disability; geotagging
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: two groups, repeated measures, pre and post intervention measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): The intervention group will be mailed a Fitbit device and provided access to the RecTech Match website. Intervention participants will receive weekly calls for the first 6 weeks, and a call every other week for the following 6 weeks (9 in total) from a health coach to discuss progress, facilitate setting physical activity goals, and help mitigate obstacles to participate in physical activity in the community. Participants will be free to access the features and resources of the website. The Fitbit data will be collected on an ongoing basis and the participants will receive daily texts asking them to rate the amount of physical activity for the day.
  Interventions: Other: RecTech Match Website
- Control (No Intervention): The control participants will not have access to the RecTech Match website; however, control participants will be directed to generic information available on the NCHPAD website, which includes the same information but is not delivered through RecTechMatch.com.

INTERVENTIONS:
Other: RecTech Match Website — Participants will have access to the Rectech Match website. These participants will receive 9 health coaching calls. Fitbit physical activity data will be collected on an ongoing basis during the intervention.
  Other Names: rectechmatch.org
  Arms: intervention

SUMMARY:
The multilevel socio-ecological barriers to physical activity experienced by people with physical disabilities cut across structures and systems, community, institutions and organizations, interpersonal, and individual levels. Several studies have attempted to understand these barriers and facilitators, but to date, no study or system has attempted to systematically resolve these multilevel barriers and capitalize on the potential facilitators that can increase access to exercise and recreation programs, services and facilities for people with disabilities.

In RecTech's previous cycle of funding, this void was addressed in a Proof of Concept product called the Activity Inclusion Mapping System (AIMS). AIMS enabled people with disabilities to quickly and precisely identify accessible and usable community-based physical activity resources and services. Based on the positive feedback received at the annual RESNA conference and from our Consumer Research Advisory Committee (CRAC) during preparation of this application, the investigators propose to develop an innovative person-centered geotagged Social Networking System (SNS) based on the social-ecological model of health.

The focus of this proposed Proof of Product project is to address multilevel barriers and facilitators associated with community-based leisure time physical activity (LTPA) using crowdsourcing principles for gathering data. The project is targeted to all people with physical disabilities.

DETAILED DESCRIPTION:
The stage of development for a RecTech Match website is a Proof of Product. The RecTech Match website will be a new online resource that will provide physical activity resources inclusive of people with disabilities. Users will be able to search for accessible opportunities for physical activity near them, watch videos on-demand related to exercise, and read articles to learn about exercise or introduce them to new community exercise opportunities. Once successful feasibility testing is completed, the investigators will work with nchpad.org, to seed information and launch nationally.

Thirty users with physical disabilities, ages 18 to 64, will participate in a 12-wk two-arm parallel randomized control trial (15 per group) aimed at reducing barriers to physical activity, increasing social support and increasing leisure-time physical activity minutes. A sample of 15 per arm will be sufficient for our pilot/feasibility study. The control arm will have access to generic information available on the National Center on Health Physical Activity and Disability (NCHPAD) website, which includes the same information but is not delivered through RecTechMatch.com. All users will be recruited online. Fitbit sensors will be provided to participants to objectively measure physical activity minutes Process feasibility outcome measures will include recruitment, retention and adherence, and Intervention efficacy outcomes will include the Godin-Shephard Leisure-Time Physical Activity Questionnaire, the Barriers to Physical Activity Questionnaire for People with Mobility Impairments (BPAQ-MI), and Chogahara's Social Influence on Physical Activity questionnaire. Daily self-report physical activity will be collected by secure email or text. Health Coaching calls and exit interviews will be recorded via Twilio Flex.

After baseline assessments are completed by all participants, each will be randomized to the 2 study arms in a 1:1 Each participant will be randomly assigned (through REDCap) to 1 of 2 treatment conditions: (1) RecTech match intervention with tele-coaching support, and (2) control. All participants will receive a welcome call and asked to provide days and times that are most convenient to attend tele-health coaching calls. Intervention group participants will receive an orientation call once shipment is received of the Fitbit device to help set the device up and ready for data collection.

The intervention group will be mailed a Fitbit device and provided access to the RecTech Match website. These participants will receive weekly calls for the first 6 weeks, and a call every other week for the following 6 weeks (9 in total) from a health coach to discuss intervention progress, facilitate setting physical activity goals, and help mitigate obstacles to participate in physical activity in the community. Participants will be free to access the features and resources of the website. The Fitbit data will be collected on an ongoing basis and the participants will receive daily texts asking them to rate the amount of physical activity for the day.

The control participants will not have access to the RecTech Match website; however, control participants will be directed to generic information available on the NCHPAD website, which includes the same information but is not delivered through RecTechMatch.com.

All participants will receive survey packets through RedCap's auto-delivery system. Survey packets will be delivered at 12 and 24 weeks. Additionally, Intervention participants will participate in a short exit interview.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 64 years old
2. self-reported physical disability that limits their mobility

Exclusion Criteria:

1. Cognitive or linguistic problems with understanding instructions or filling in self-administered outcome measures
2. Cardiovascular disease event within the past 6 months
3. Severe pulmonary disease or renal failure
4. Currently pregnant
5. Ongoing exacerbation of a health condition
6. Other conditions that would interfere with being physically active

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Godin - Leisure time physical activity questionnaire | pre-intervention and again at the end of 12 weeks
  Estimates habitual leisure time physical activity. Higher numbers indicate more times the person has engaged in physical activity separated by 3 categories. There is no scoring limit.
Barriers to Physical Activity Questionnaire for People with Mobility Impairments | pre-intervention and again at the end of 12 weeks
  Identifies barriers to physical activity, specifically designed for individuals with a mobility. impairment. The survey has 8 subscales (health, beliefs and attitudes, family, friends, fitness-center-built environment, staff and policy, community built environment, and safety. Subscale scores of 1 to 5 are calculated. Higher values indicate a higher influence of barriers.
Chogahara's Social Influence on Physical Activity Questionnaire | pre-intervention and again at the end of 12 weeks
  Measures a persons perceptions on how their physical activity is affected by social influences. The survey has 3 factors (friends, family, and health/fitness expert) and 3 subscales (companionship, informational, and emotional support). Each subscale can have a minimum maximum score of 4 with a higher score indicating a higher frequency of influence.
Post Intervention Interviews | pre-intervention and again at the end of 12 weeks
  Gather feedback on the end user's experiences using the website.

SECONDARY OUTCOMES:
FitBit device data (total energy expenditure, steps, sedentary time, light activity time, moderate activity time, high activity time, and activity energy expenditure). | FitBit Data will be continuously collected for 12 weeks
  The Fitbit device reports, the total amount of energy expended (kCal) per day, the number of steps achieved per day, the number of minutes that the wearer engaged either sedentary activity or physical activity (light, moderate, high), and finally the energy expenditure cost of the physical activity (kCAL) per day.

CONTACTS AND LOCATIONS:
Locations (1):
- UAB / Lakeshore Research Collaborative, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martin Ginis KA, Ma JK, Latimer-Cheung AE, Rimmer JH. A systematic review of review articles addressing factors related to physical activity participation among children and adults with physical disabilities. Health Psychol Rev. 2016 Dec;10(4):478-494. doi: 10.1080/17437199.2016.1198240. Epub 2016 Jun 29. PMID 27265062
- [Background] Vasudevan V, Rimmer JH, Kviz F. Development of the Barriers to Physical Activity Questionnaire for People with Mobility Impairments. Disabil Health J. 2015 Oct;8(4):547-56. doi: 10.1016/j.dhjo.2015.04.007. Epub 2015 May 14. PMID 26087721
- [Background] McLeroy KR, Bibeau D, Steckler A, Glanz K. An ecological perspective on health promotion programs. Health Educ Q. 1988 Winter;15(4):351-77. doi: 10.1177/109019818801500401. PMID 3068205
- [Background] Takacs J, Pollock CL, Guenther JR, Bahar M, Napier C, Hunt MA. Validation of the Fitbit One activity monitor device during treadmill walking. J Sci Med Sport. 2014 Sep;17(5):496-500. doi: 10.1016/j.jsams.2013.10.241. Epub 2013 Oct 31. PMID 24268570
- [Background] Amireault S, Godin G. The Godin-Shephard leisure-time physical activity questionnaire: validity evidence supporting its use for classifying healthy adults into active and insufficiently active categories. Percept Mot Skills. 2015 Apr;120(2):604-22. doi: 10.2466/03.27.PMS.120v19x7. Epub 2015 Mar 23. PMID 25799030
- [Background] Chogahara M. A multidimensional scale for assessing positive and negative social influences on physical activity in older adults. J Gerontol B Psychol Sci Soc Sci. 1999 Nov;54(6):S356-67. doi: 10.1093/geronb/54b.6.s356. PMID 10625971
- See also: The National Center on Health, Physical Activity, and Disability — https://www.nchpad.org/